CLINICAL TRIAL: NCT01048983
Title: A Study of Reducing the Symptom Burden Produced by Chemoradiation Treatment for Non Small Cell Lung Cancer
Brief Title: Reducing Symptom Burden - Non Small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2008-0345; R01 026582-26 (Other: NCI); NCI-2012-01256 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer; NSCLC; Concurrent Chemoradiation Therapy; Side Effects; Armodafinil; Nuvigil; Bupropion; Wellbutrin; Wellbutrin SR; Zyban; Curcumin; Minocycline; Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; cyclopia sequence | interventions — Modafinil; Bupropion; Minocycline; Curcumin; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (16):
- Questionnaires and Phone Calls (Other): Weeks 1-10, 2 questionnaire calls/week; and Weeks 11-16, 1 call/week.
  Interventions: Behavioral: Telephone Questionnaire
- Curcumin Only (Active Comparator)
  Interventions: Drug: Curcumin; Behavioral: Telephone Questionnaire
- Armodafinil Only (Active Comparator)
  Interventions: Drug: Armodafinil; Behavioral: Telephone Questionnaire
- Minocycline Only (Active Comparator)
  Interventions: Drug: Minocycline; Behavioral: Telephone Questionnaire
- Bupropion Only (Active Comparator)
  Interventions: Drug: Bupropion; Behavioral: Telephone Questionnaire
- Curcumin + Armodafinil (Active Comparator)
  Interventions: Drug: Armodafinil; Drug: Curcumin; Behavioral: Telephone Questionnaire
- Curcumin + Minocycline (Active Comparator)
  Interventions: Drug: Minocycline; Drug: Curcumin; Behavioral: Telephone Questionnaire
- Curcumin + Bupropion (Active Comparator)
  Interventions: Drug: Bupropion; Drug: Curcumin; Behavioral: Telephone Questionnaire
- Armodafinil + Minocycline (Active Comparator)
  Interventions: Drug: Armodafinil; Drug: Minocycline; Behavioral: Telephone Questionnaire
- Armodafinil + Bupropion (Active Comparator)
  Interventions: Drug: Armodafinil; Drug: Bupropion; Behavioral: Telephone Questionnaire
- Minocycline + Buproprion (Active Comparator)
  Interventions: Drug: Bupropion; Drug: Minocycline; Behavioral: Telephone Questionnaire
- Curcumin + Armodafinil + Minocycline (Active Comparator)
  Interventions: Drug: Armodafinil; Drug: Minocycline; Drug: Curcumin; Behavioral: Telephone Questionnaire
- Curcumin + Armodafinil + Bupropion (Active Comparator)
  Interventions: Drug: Armodafinil; Drug: Bupropion; Drug: Curcumin; Behavioral: Telephone Questionnaire
- Curcumin + Minocycline + Bupropion (Active Comparator)
  Interventions: Drug: Bupropion; Drug: Minocycline; Drug: Curcumin; Behavioral: Telephone Questionnaire
- Armodafinil + Minocycline + Bupropion (Active Comparator)
  Interventions: Drug: Armodafinil; Drug: Bupropion; Drug: Minocycline; Behavioral: Telephone Questionnaire
- Curcumin + Armodafinil + Minocycline + Bupropion (Active Comparator)
  Interventions: Drug: Armodafinil; Drug: Bupropion; Drug: Minocycline; Drug: Curcumin; Behavioral: Telephone Questionnaire

INTERVENTIONS:
Drug: Armodafinil — Initial Dose 150 mg once a day (50 mg and 100 mg oral tablets) for 10 weeks.
  Other Names: Nuvigil; Modafinil
  Arms: Armodafinil + Bupropion; Armodafinil + Minocycline; Armodafinil + Minocycline + Bupropion; Armodafinil Only; Curcumin + Armodafinil; Curcumin + Armodafinil + Bupropion; Curcumin + Armodafinil + Minocycline; Curcumin + Armodafinil + Minocycline + Bupropion
Drug: Bupropion — Initial Dose 100 mg two times a day (200 mg) for 10 weeks.
  Other Names: Wellbutrin; Wellbutrin SR; Zyban
  Arms: Armodafinil + Bupropion; Armodafinil + Minocycline + Bupropion; Bupropion Only; Curcumin + Armodafinil + Bupropion; Curcumin + Armodafinil + Minocycline + Bupropion; Curcumin + Bupropion; Curcumin + Minocycline + Bupropion; Minocycline + Buproprion
Drug: Minocycline — Initial Dose 100 mg two times a day (200 mg) for 10 weeks.
  Other Names: Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
  Arms: Armodafinil + Minocycline; Armodafinil + Minocycline + Bupropion; Curcumin + Armodafinil + Minocycline; Curcumin + Armodafinil + Minocycline + Bupropion; Curcumin + Minocycline; Curcumin + Minocycline + Bupropion; Minocycline + Buproprion; Minocycline Only
Drug: Curcumin — Initial Dose 4 gm stick pack once a day (4 gm) for 10 weeks.
  Arms: Curcumin + Armodafinil; Curcumin + Armodafinil + Bupropion; Curcumin + Armodafinil + Minocycline; Curcumin + Armodafinil + Minocycline + Bupropion; Curcumin + Bupropion; Curcumin + Minocycline; Curcumin + Minocycline + Bupropion; Curcumin Only
Behavioral: Telephone Questionnaire — Weeks 1-10, 2 questionnaire calls/week; and Weeks 11-16, 1 call/week.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to compare armodafinil, bupropion, curcumin, and minocycline when given alone or in combination to learn which is better for controlling symptoms, such as the side effects of chemoradiation, when given to treat lung cancer.

DETAILED DESCRIPTION:
The Study Drugs:

It is not known which study drug or combination of study drugs is better at reducing side effects patients may experience during chemoradiation therapy. For this reason, researchers have chosen 4 study drugs that may help to reduce side effects. The study drugs will be tested alone and in combination with each other.

Armodafinil is designed to prevent excessive sleepiness.

Bupropion is an antidepressant with anti-inflammatory properties that may help reduce multiple symptoms.

Curcumin is the active ingredient in the spice, turmeric. It may interfere with the production of cytokines (which cause inflammation), which may reduce multiple symptoms.

Minocycline is an antibiotic. Minocycline has been shown to interrupt cytokine production, which may help to reduce multiple symptoms.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the roll of dice) to join 1 of 16 groups. You may be assigned to receive no study drugs, 1 study drug, or a combination of 2, 3, or all 4 of the study drugs.

During this study, you may receive 1 or more placebos. A placebo looks like the study drug(s) but has no active ingredients. There is a chance that you will be in a group that does not receive any study drugs at all. However, all patients are under standard care by their treating doctors.

Neither you nor the study staff you will see in the clinic will know if you are receiving the study drugs and/or the placebo(s). However, if needed for your safety, the study staff will be able to find out which study drug you are receiving.

Study Drug Administration:

You will take the study drugs/placebos every day for 10 weeks. You will take either single or combined study drug(s) or placebos by mouth everyday as instructed by the study doctor.

You will be given pamphlets with more information about how to take the study drugs/placebos.

You will be given a daily diary to write down when you take the study drugs/placebo. You should bring your study drug/placebo blister packs/sticks to the clinic to every study visit. You should also bring your diary to every visit.

Completing the Symptom Questionnaire:

Throughout the study, you will be asked to complete the symptom questionnaire. You will be asked about symptoms from therapy you may be experiencing and how they may be interfering with your daily activities. The study staff will either meet you during your regular clinic visit or call you at your home at a time that is convenient for you. In the clinic, you will complete the questionnaire by paper and pen, or by entering your answers into an electronic tablet computer. On the phone, study staff will ask you the questions and record your answers on paper or enter them into a computer. The symptom questionnaire will take up to 5 minutes to complete.

* During Weeks 1-10, you will complete the symptom questionnaire 2 times a week.
* During Weeks 11-16, you will complete the symptom questionnaire 1 time a week.

Study Visits:

Before you begin chemoradiation:

* You will complete 4 questionnaires about pain and other symptoms, your mood, and your quality of life. Completing all 4 of the questionnaires will take about 15 minutes.
* You will have a blood coagulation test, called a PT-INR, to make sure your blood clots normally.
* If you are a woman who is able to become pregnant, you will have a urine pregnancy test. The study staff will give you the pregnancy test kit at your scheduled visit, and will review and record the results of the test before your study prescriptions are filled by the pharmacy.

After 4 weeks of chemoradiation:

* You will complete 1 questionnaire about your quality of life. This questionnaire will take about 2-3 minutes to complete.
* You will have a blood coagulation test, called a PT-INR, to make sure your blood clots normally.

During the last week of chemoradiation (about Week 7):

-You will complete 3 questionnaires about your symptoms, mood, and quality of life. These questionnaires will take about 10 minutes total to complete.

After about Week 7, the study staff will call you 2 times a week to check on you until week 10. This phone call should last only a few minutes. If you have experienced several side effects from chemoradiation, this phone call make take longer.

About Week 12 (at a routine clinical visit):

* You will complete 3 questionnaires about your symptoms, mood, and quality of life.
* If you were smoking at the beginning of the study, you will complete a questionnaire that asks if you stopped smoking any time during the study. This will take a few minutes.
* You will have a blood coagulation test, called a PT-INR, to make sure your blood clots normally.
* You will be asked to complete another questionnaire that asks about your satisfaction with the study drug(s). This will take a few minutes.

Length of Study:

You will be on study for about 16 weeks. You will take the study drug(s) for 10 weeks and complete the symptom survey until 16 weeks. You will be taken off study if you experience intolerable side effects.

This is an investigational study. Armodafinil is FDA approved and commercially available for the treatment of excessive sleepiness. Bupropion is FDA approved and commercially available for the treatment of depression. Minocycline is FDA approved and commercially available for the treatment of bacterial infection. Curcumin is not FDA approved. At this time, curcumin is only being used in research. The different possible combinations of these drugs being used in this study is investigational.

Up to 32 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathologically proven diagnosis of unresectable Non-small-cell lung carcinoma (NSCLC) and consented to concurrent chemoradiation therapy in MD Anderson Cancer Center (MDACC).
2. Patients >= 18 years old and <= 65 years old
3. Patients who will receive chemoradiation with platinum/taxane based chemo and with a total radiation dose of > or = 50 Gy, per treating physician's assessment
4. Patients who speak English only (due to the novel research and its complexity, we are only accruing English speaking patients to the protocol)
5. Patients must agree to discontinue any current herbal supplement use, and refrain from taking any herbal supplement while on protocol
6. Patients must be willing and able to review, understand, and provide written consent before starting therapy
7. Patients already taking any of this trial's symptom treatment medications (including modafinil) must be willing to stop taking the medication/s for a washout period of 30 days before they are randomized to a symptom treatment arm and begin the symptom trial

Exclusion Criteria:

1. Patients who are taking medications or have conditions that potentially preclude use of any study medications or interventions as determined by the treating physician
2. Patients taking CHANTIX (smoking cessation medication)
3. Patients who are enrolled in other symptom management or treatment clinical trials
4. Bile duct obstruction or cholelithiasis
5. History of clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, including multiple allergies or drug reaction
6. Pre-existing psychosis or bipolar disorder
7. Pre-existing renal impairment: The screening cut off for serum creatinine >1.5mg/dl will be done by the oncologist to qualify for CXRT.
8. Pre-existing hepatic impairment: The screening for total bilirubin >25.7 µmol/L (1.5 mg/dL) will be done by the oncologist to qualify for chemoradiation treatment (CXRT). The screening for 2 times the upper limit of normal Hepatotoxicity (Aspartate aminotransferase (AST), Alkaline phosphatase (ALP) and Alanine aminotransferase (ALT) will be done by the oncologist to qualify for CXRT.
9. Pre-existing Tourette's syndrome
10. Seizure disorder
11. Anorexia/bulimia in past two months
12. Use of monoamine oxidase (MAO) inhibitors within 14 days
13. Patients undergoing abrupt discontinuation of ethanol or sedatives (including benzodiazepines)
14. Patients receiving other dosage forms of bupropion if they do not agree to undergo a washout period
15. Allergy to turmeric or any of its constituents, including curcumin, to yellow food coloring, or to member of the Zingiberaceae (ginger) family
16. Gastric or duodenal ulcers, or gastric hyperacidity disorders
17. Hypersensitivity to any tetracyclines
18. Patients to be confirmed as not pregnant (serum HCG negative). The screening for this will be done by the oncologist in qualifying for CXRT.
19. Patients with a history of cardiac disease, including angina and cardiac ischemia, left ventricular hypertrophy, myocardial infarction, and mitral valve prolapse.
20. Patients taking antifungals, antiretrovirals, and macrolides that are strong CYP3A4 strong inhibitors including indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, and nefazodone.
21. Patients on anticoagulants (ie warfarin/heparin)
22. Patients with International Normalized Ratio (INR) > 1.5.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Combined AUC for Selected Symptoms | 10-weeks (+/- 4 days)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongxing Liao, MD, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org